CLINICAL TRIAL: NCT00337415
Title: Proprietary Information - Exploratory (Non-Confirmatory) Trial
Brief Title: MK0354 Clinical Efficacy and Tolerability Study (0354-004)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0354-004
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — 3-(1H-tetrazol-5-yl)-1,4,5,6-tetrahydrocyclopentapyrazole

INTERVENTIONS:
Drug: MK0354

SUMMARY:
A Research Study to Evaluate the Effectiveness and Tolerability of MK0354 vs Placebo (an inactive look alike pill) in Lipid (fat) Altering in Patients with dyslipidemia (a disorder of lipids in the blood)

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age
* You have taken a statin or other lipid modifying therapy in the last 6-8 weeks
* You have lipid lab values outside of the range specified in the protocol

Exclusion Criteria:

* Patient is a woman who is pregnant or nursing a child
* Patient is a woman who is taking hormonal birth-control
* You are a woman who is planning to donate eggs during the study
* You plan to give blood during the study or have given within the last 8 weeks
* You are a woman who is having menopausal hot flashes or are taking medications to prevent menopausal hot flashes
* You have a known intolerance to or you are allergic to niacin
* You have any of the following medical conditions:
* Poorly controlled or newly diagnosed diabetes (within the last 3 months)
* Thyroid disease (hypothyroidism or hyperthyroidism)
* A history of stroke, heart attack, coronary bypass surgery, angioplasty, unstable angina or similar heart and artery procedures in the past 3 months
* History of hemorrhagic stroke or other non-traumatic hemorrhage
* Peptic ulcer disease in the last 3 months
* An occurrence of gout within the last year and you are not currently taking allopurinol
* Cancer (except for successfully treated skin cancer)
* HIV positive
* You have a history of drug/alcohol abuse within the last year
* You consume more than 2 drinks of alcohol per day
* You do not have access to a telephone
* You take medications that are not allowed in this study. The study doctor or staff will discuss this with you.
* Patient has participated in a study with an investigational drug within the last 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
proprietary information - exploratory (non-confirmatory) trial

SECONDARY OUTCOMES:
proprietary information - exploratory (non-confirmatory) trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC